CLINICAL TRIAL: NCT04396197
Title: Physical Activity Levels in COVID-19 Patients Admitted to Intensive Care Requiring Invasive Ventilation: An Observational Study
Brief Title: Physical Activity Levels in COVID-19 Patients Admitted to Intensive Care
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David McWilliams, Consultant Physiotherapist, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: PhysioCOVID-19
Record Dates: First submitted 2020-05-17; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Critical Illness; Ards; ICU Acquired Weakness
MeSH Terms: conditions — COVID-19; Critical Illness; Acute Lung Injury | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Observations taken of standard physiotherapy practice. All patients are assessed daily and receive respiratory care and rehabilitation as deemed appropriate by the treating therapist
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Daily physiotherapy to include respiratory care and rehabilitation based on the individual therapists clinical reasoning
  Other Names: Rehabilitation

SUMMARY:
This is an observational study exploring the levels of mobility and rehabilitation in patients admitted to critical care with a confirmed diagnosis of COVID-19

DETAILED DESCRIPTION:
An admission to an intensive care unit (ICU) often results in significant muscle weakness and physical deconditioning, which can take many months or even years for recovery. Early and progressive programmes of rehabilitation are recommended to limit any muscle loss and support recovery as early as possible. Patients admitted to intensive care with COVID-19 have been found to require prolonged periods of mechanical ventilation, high sedation and neuromuscular blocking use and as a result require prolonged stays in the ICU. As yet no data exists to examine the specific physical impact this may have, or whether it is safe and feasible to commence this earlier rehabilitation within the ICU for patients with a diagnosis of COVID-19. Our study set out to evaluate the levels of rehabilitation which were delivered in a large acute NHS trust.

ELIGIBILITY:
Inclusion Criteria:

* having a confirmed diagnosis of COVID-19
* being mechanically ventilated for at least 24 hours
* surviving to critical care discharge.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults admitted to ICU with a confirmed diagnosis of COVID-19, mechanically ventilated for >24 hours and surviving to ICU discharge were included.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
Mobility level | At ICU discharge, an average of 3 weeks
  Highest level of mobility achieved at the point of ICU discharge
Time taken to first mobilise | during ICU admission, up to 3 weeks
  Time taken to first mobilise, defined as sitting on the edge of the bed or higher

SECONDARY OUTCOMES:
Discharge location | Hospital discharge, up to 2 months
  Discharged to home, home with rehab, or a community rehab facility

CONTACTS AND LOCATIONS:
Locations (1):
- UHB NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McWilliams D, Weblin J, Hodson J, Veenith T, Whitehouse T, Snelson C. Rehabilitation Levels in Patients with COVID-19 Admitted to Intensive Care Requiring Invasive Ventilation. An Observational Study. Ann Am Thorac Soc. 2021 Jan;18(1):122-129. doi: 10.1513/AnnalsATS.202005-560OC. PMID 32915072